CLINICAL TRIAL: NCT04286776
Title: Memory Retrieval and Encoding Investigated by Neural Stimulation
Acronym: MEMREINS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 820553; 1U01NS113198-01 (NIH); 5R01NS106611-05 (NIH)
Record Dates: First submitted 2020-02-24; First posted 2020-02-27 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Epilepsy Intractable
Keywords: episodic memory
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: All enrolled patients are considered eligible to receive direct electrical stimulation. Subjects have the option to receive non stimulation testing only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Direct Electrical Stimulation (Experimental): Stimulation will be applied concurrently with the task, if applicable, and stimulation trials will be interleaved with sham trials, where no stimulation is delivered.
  Interventions: Device: Direct electrical stimulation

INTERVENTIONS:
Device: Direct electrical stimulation — Stimulation will not exceed 0.75 mA and will be approved prior by study investigators. Each subject will have a safety threshold testing at the beginning of each session and if 'afterdischarges' occur the subject's stimulation threshold will be lowered.

SUMMARY:
The purpose of this research is to understand biomarkers of human memory through correlational analyses and to use focal electrical stimulation as a causal manipulation to understand how biomarkers of memory relate to other brain states and behavioral measures.

ELIGIBILITY:
Inclusion Criteria:

1. Expected to undergo intracranial implantation and postoperative electroencephalographic monitoring as part of a standard clinical procedure for the treatment of pharmacologically resistant epilepsy
2. Age 18 or older

Exclusion Criteria:

1. Any physical or cognitive disability or illness that would limit their ability to perform cognitive tasks
2. Any medical condition that would, in the investigator's opinion, limit the subject's participation in the study.
3. Unable or unwilling to provide informed consent
4. MRI contraindications

Standard clinical care includes a pregnancy test for female patients prior to the surgical implantation of the electrodes. Pregnant women are not surgically implanted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2014-10-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To use direct electrical stimulation to disentangle causal versus correlative biomarkers of verbal and spatial episodic memory | Up to 4 weeks (typical duration of hospital stay)
  1. We will use linear mixed effects models and L2-penalized logistic regression classifiers to compare periods of successful and unsuccessful performance in our tasks
To develop and test models of human brain dynamics in the presence of electrical stimulation | Up to 4 weeks (typical duration of hospital stay)
  2. We will compare spectral indices of brain activity before and after stimulation as a function of stimulation parameters.
To assess how reactivation of prior memories shapes subsequent recall and memory organization, including memory for the content, context and value of experiences. | Up to 4 weeks (typical duration of hospital stay)
  3. We will mathematical models of neural similarity described in detail in Halpern (2024) and Manning (2011, 2012) to test the reactivation mechanisms described in Lohnas et al. (2014) and Healey and Kahana (2015).
To determine whether state-dependent stimulation can separately be used to modulate encoding and retrieval processes | Up to 4 weeks (typical duration of hospital stay)
  4. We will evaluate the closed-loop stimulation protocol described in Kahana et al. (2023) in both encoding and retrieval.
To determine whether stimulation is more effective at modulating memory when targeted to regions with specific connectivity profiles to the medial temporal lobe | Up to 4 weeks (typical duration of hospital stay)
  5. We will compare recall rates during a free recall experiment with brain stimulation at sites with high network-mediated activation, as described in Solomon et al. (2018), versus low network-mediated activation.
To determine how simultaneous stimulation at multiple target sites can be optimized to modulate memory | Up to 4 weeks (typical duration of hospital stay)
  6. We will compare recall rates during a free recall experiment with no brain stimulation, stimulation at one site, and stimulation at multiple sites.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kahana, PhD, Principal Investigator — University of Pennsylvania
Locations (11):
- United States (11):
  - University of Colorado, Denver, Aurora, Colorado
  - Emory University Hospital, Atlanta, Georgia
  - National Institute of Neurological Disorders and Stroke, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared in a public repository at regular intervals during the project. De-identified data sets will be anonymized prior to posting on the public repository. These de-identified data are likely to be analyzed for secondary purposes other than those described in this protocol (e.g. seizure prediction). Shared data will include, at a minimum, digital spreadsheets used to summarize all participant behavioral data. De-identified electrophysiology data, demographic information, electrode localization information, and task information (e.g. timing of each trial, timing of responses) will be shared in a central repository. Descriptions of the tasks and stimuli will be shared. De-identified references to individual participant data may also appear in scientific journal publications or presented at scientific meetings.
Time Frame: Study data will become available within six months of publication of the relevant results, with no planned expiration.
Access Criteria: Data is freely available, will require a formal request for access.

REFERENCES:
- [Background] Ezzyat Y, Kragel JE, Solomon EA, Lega BC, Aronson JP, Jobst BC, Gross RE, Sperling MR, Worrell GA, Sheth SA, Wanda PA, Rizzuto DS, Kahana MJ. Functional and anatomical connectivity predict brain stimulation's mnemonic effects. bioRxiv [Preprint]. 2023 Aug 11:2023.07.27.550851. doi: 10.1101/2023.07.27.550851. PMID 37609181
- [Background] Ezzyat Y, Wanda PA, Levy DF, Kadel A, Aka A, Pedisich I, Sperling MR, Sharan AD, Lega BC, Burks A, Gross RE, Inman CS, Jobst BC, Gorenstein MA, Davis KA, Worrell GA, Kucewicz MT, Stein JM, Gorniak R, Das SR, Rizzuto DS, Kahana MJ. Closed-loop stimulation of temporal cortex rescues functional networks and improves memory. Nat Commun. 2018 Feb 6;9(1):365. doi: 10.1038/s41467-017-02753-0. PMID 29410414
- [Background] Kragel JE, Ezzyat Y, Lega BC, Sperling MR, Worrell GA, Gross RE, Jobst BC, Sheth SA, Zaghloul KA, Stein JM, Kahana MJ. Distinct cortical systems reinstate the content and context of episodic memories. Nat Commun. 2021 Jul 21;12(1):4444. doi: 10.1038/s41467-021-24393-1. PMID 34290240